CLINICAL TRIAL: NCT00258232
Title: Phase II Study of Celecoxib, Capecitabine, and Irinotecan in Patients With Metastatic Colorectal Cancer
Brief Title: Celecoxib, Capecitabine, and Irinotecan in Treating Patients With Recurrent or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445439; P30CA022453 (NIH); WSU-C-2424
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; recurrent rectal cancer; stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Celecoxib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine
Drug: celecoxib
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as capecitabine and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving celecoxib together with capecitabine and irinotecan may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving celecoxib together with capecitabine and irinotecan works in treating patients with recurrent or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with locally recurrent or metastatic colorectal cancer treated with celecoxib, capecitabine, and irinotecan.

Secondary

* Determine the time to progression in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the overall survival of patients treated with this regimen.
* Determine the time to treatment failure in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral celecoxib twice daily on days -7 to 21 during course 1 and on days 1-21 in all subsequent courses. Patients also receive oral capecitabine twice daily on days 1-14 and irinotecan IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete or partial response after 4 courses may temporarily discontinue treatment for no more than 4 weeks.

After completion of study treatment, patients are followed every 6 months for survival.

PROJECTED ACCRUAL: A total of 21-44 patients will be accrued for this study within 7-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Locally recurrent or metastatic disease
* Measurable disease, defined as ≥ 1 measurable lesion ≥ 20 mm by conventional CT scan OR ≥ 10 mm by spiral CT scan

  * Bone metastases, ascites, and pleural effusion are not considered measurable disease
  * Measurable lesions must be located outside a previously irradiated field

PATIENT CHARACTERISTICS:

Performance status

* SWOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* No Gilbert's disease

Renal

* Creatinine clearance > 50 mL/min

Cardiovascular

* No clinically significant cardiac disease that is not well controlled by medication, including any of the following conditions:

  * Congestive heart failure
  * Symptomatic coronary artery disease
  * Cardiac arrhythmias
* No myocardial infarction within the past year

Gastrointestinal

* Must have a physically intact upper gastrointestinal tract
* Able to swallow tablets
* No history of peptic ulcer disease or gastroesophageal reflux
* No malabsorption syndrome

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* No asthma, urticaria, or allergic-type reaction after prior treatment with aspirin or other nonsteroidal anti-inflammatory drugs
* No other malignancy except curatively treated cancer with no evidence of active disease
* No unresolved bacterial infection requiring antibiotics
* No other serious infection
* No known allergy to study drugs or sulfa drugs

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for colorectal cancer

  * Patients relapsing > 6 months after completion of prior adjuvant chemotherapy allowed
* No other concurrent anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy
* No concurrent anticancer radiotherapy

Surgery

* Recovered from prior surgery
* No concurrent anticancer surgery

Other

* Prior celecoxib for nonmalignant disorders allowed
* No other concurrent cyclooxygenase-2 inhibitors or nonsteroidal anti-inflammatory drugs, including any of the following:

  * Rofecoxib
  * Ibuprofen
  * Naproxen
  * Etodolac
  * Oxaprozin
  * Diflunisal
  * Nabumetone
  * Tolmetin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2007-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Response rate by RECIST criteria at every other course

SECONDARY OUTCOMES:
Time to progression
Toxicity
Overall survival
Time to treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, MD, PhD, FRCP, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (3):
- United States (3):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] El-Rayes BF, Venkat R, Heilbrun LK: A dose attenuated schedule of irinotecan and capecitabine in combination with celecoxib in advanced colorectal cancer. [Abstract] American Society of Clinical Oncology 2006 Gastrointestinal Cancers Symposium, 26-28 January 2006, San Francisco, California. A-254, 2006.